CLINICAL TRIAL: NCT00993720
Title: Effect of GLP-1 on Insulin-dose, Risk of Hypoglycemia and Gastric Emptying Rate in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Sten Madsbad, MD, chief physician, Hvidovre University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-001930-80
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus
Keywords: patients with type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- type 1 DM with betacell function: Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- type 1 DM without betacell function: Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- type 1 DM without betacell function: Insulin (No Intervention)
  Interventions: Other: continuous insulin therapy

INTERVENTIONS:
Drug: Liraglutide — after optimal treatment on insulin alone 10 patients with type 1 diabetes are treated for four weeks with Liraglutide : in the first week at 0.6 mg sc and after one week optitration to the recommended 1.2 mg sc pr day.
  Arms: type 1 DM with betacell function: Liraglutide
Drug: Liraglutide — after optimal treatment with insulin alone, 10 type 1 diabetic patients are treated with Liraglutide at a dose of 0.6 mg sc. After one week the dose is optitreted to the recommended 1.2 mg sc pr. day.
  Arms: type 1 DM without betacell function: Liraglutide
Other: continuous insulin therapy — after optimal treatment with insulin, patients continue on insulin for four weeks
  Arms: type 1 DM without betacell function: Insulin

SUMMARY:
The aim of the study is to investigate the effect of Victoza (a GLP-1 receptor agonist)on insulin-dose, risk of hypoglycemia and gastric emptying rate during hypoglycemia in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50y,
* BMI 18-27,
* caucasian origin,
* type 1 diabetes diagnosed between age 5 and age 40,
* no known diabetes complications or cardiovascular diseases,
* no medication known to influence glucose homeostasis,
* no pregnancy

Exclusion Criteria:

* diabetes complications,
* autonomous nerve dysfunction,
* anaemia,
* HbA1c < 8.5% at screening,
* estimated by the investigator to be incapable of completing the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
insulin-dose | 4 weeks

SECONDARY OUTCOMES:
24-hours glucose profiles with and without treatment of Victoza | three days
risk of hypoglycemia during physical activity with and without Victoza | one day
gastric emptying rate during hypoglycemia with and without Victoza | one day
weight change from baseline, change in fructosamine from baseline | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Kielgast U, Krarup T, Holst JJ, Madsbad S. Four weeks of treatment with liraglutide reduces insulin dose without loss of glycemic control in type 1 diabetic patients with and without residual beta-cell function. Diabetes Care. 2011 Jul;34(7):1463-8. doi: 10.2337/dc11-0096. Epub 2011 May 18. PMID 21593296